CLINICAL TRIAL: NCT05031000
Title: Cheap Equals Bad? Comparative System Accuracy of POCT Blood Glucose Monitoring Systems Under the Aspect of Aspect of Pricing: Discounter Versus Brand
Brief Title: Blood Glucose Monitoring Systems: Discounter Versus Brand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDK_ISO_2021_002
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject POCT glucometer measurement (Experimental): Blood glucose measurement POCT glucometer
  Interventions: Diagnostic Test: blood glucose measurement: POCT; Diagnostic Test: blood glucose measurement: reference

INTERVENTIONS:
Diagnostic Test: blood glucose measurement: POCT — measurement of blood glucose concentration using 5 different POCT glucometer
Diagnostic Test: blood glucose measurement: reference — measurement of blood glucose concentration using 2 different laboratory analyzer

SUMMARY:
This study assesses the system accuracy of 5 blood glucose monitoring systems pursuant to ISO 15197 under the aspect of the system's prospected costs for the user.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with clinical indication for blood glucose measurement
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with inherent risk of aggravation by the procedure (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* A current constitution that does not allow participating in the study (e.g. hematocrit out of BGM specifications, medication known to influence blood glucose measurements; see Appendix A of ISO 15197)
* Being unable to give informed consent
* < 18 years
* Legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Analysis of system accuracy based on DIN EN ISO 15197 | day 1
  Assessment of the analytical measurement performance of 5 blood glucose montoring systems based on procedures defined in DIN EN ISO 15197

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Salzsieder, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Blood sugar — https://medlineplus.gov/bloodsugar.html
- See also: ISO 15197 — https://www.iso.org/standard/54976.html